CLINICAL TRIAL: NCT03402529
Title: Added Value of Contrast Enhanced Spectral Mammography, CESM in Diagnostics and Size Estimation of Malignant Lesions in Breast. A Pilot Study.
Brief Title: Added Value of Contrast Enhanced Spectral Mammography, CESM. A Pilot Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/505
Record Dates: First submitted 2017-12-04; First posted 2018-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
Keywords: Contrast Enhanced Spectral Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CESM (Other)
  Interventions: Diagnostic Test: Contrast Enhanced Spectral Mammography

INTERVENTIONS:
Diagnostic Test: Contrast Enhanced Spectral Mammography — Pilot study

SUMMARY:
Introduction: To avoid unnecessary mastectomies and reoperations a correct size assessment of malignant lesions in breast is required. Sometimes a supplementary MRI is therefore recommended. However, at our unit MRI is not easily available. Contrast enhanced spectral mammography (CESM) has in smaller studies been shown to be equal to MRI regarding sensitivity and specificity. Size assessment using contrast-based modalities as CESM has also been shown to be significantly more accurate than using mammography. Prospective randomized studies using CESM are lacking.

Aim: The aim of the study is to evaluate the added value of CESM in diagnostics of breast cancer and choice of operation; partial mastectomy or mastectomy.

A pilot study of 50 patients will be conducted to prepare for a larger prospective randomized study.

Method: Patients found with breast cancer after diagnostics with mammography, ultrasound and core biopsy, and whom are recommended primary surgery, will be enrolled in the study. A supplementary examination with CESM will be performed. Preoperative extent of the malignant lesions are estimated with each modality and is later compared with the extent measured in post-operative PAD. Data on weight, length, age at menopaus, use of contraceptive pills, HRT or endocrine therapy, breast volume and density is collected, as well as data of diagnosis (ductal or lobular carcinoma), surrounding DCIS, histological grade, ER, PgR, Her2 expression and Ki67 index.

In this pilot study sensitivity and specificity for each modality is calculated. Multivariate analysis will be performed regarding influential factors. Pearson correlation coefficient will be calculated for each modality regarding size assessment of the malignant lesions in comparison with definitive PAD.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with breast cancer and whom are planned for primary surgery
* Signed informed consent

Exclusion Criteria:

* Ongoing pregnancy
* Ongoing lactation
* Allergy against iodine contrast
* Treatment with metformin (against diabetes)
* Renal failure
* Hyperthyroidism
* Severe heart condition
* Myasthenia gravis
* Implants
* Inability to understand study information

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Most breast cancers occur in women. Male breast parenchyma is very small. Not suitable to examine by contrast enhanced spectral mammography in this study
Enrollment: 47 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with change of treatment | 1 month
  Mastectomy instead of partial mastectomy, neo-adjuvant chemotherapy instead of primary surgery

SECONDARY OUTCOMES:
size assessment of malignant lesions | 2 months
  correlation with definitive PAD

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahsberg K, Gardfjell A, Nimeus E, Rasmussen R, Behmer C, Zackrisson S, Ryden L. Added value of contrast-enhanced mammography (CEM) in staging of malignant breast lesions-a feasibility study. World J Surg Oncol. 2020 May 21;18(1):100. doi: 10.1186/s12957-020-01865-0. PMID 32438917